CLINICAL TRIAL: NCT05761652
Title: An Early Warning Model for Assessing the Onset, Progression and Sequelae of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing YouAn Hospital (Other); Kossamak Hospital (Unknown); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2023XLA003-2
Record Dates: First submitted 2023-03-08; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: Early Warning Model
MeSH Terms: conditions — COVID-19 | interventions — Records

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modeling group
  Interventions: Other: Observe and record
- Validation group
  Interventions: Other: Observe and record

INTERVENTIONS:
Other: Observe and record — The general information, environmental indicators, and auxiliary examination indicators of the subjects were observed and recorded, as well as the TCM physical assessment was performed.

SUMMARY:
Based on the characteristics of symptoms, differences in physical and chemical examinations and tests, and characteristics of traditional Chinese medicine (TCM) disease differentiation and syndrome differentiation, the evaluation indicators for the clinical early warning model were screened, and the "three-level early warning mechanism for COVID-19 patients at high risks, with progression to severe cases and sequelae was constructed.

DETAILED DESCRIPTION:
Adopt multi-level evidence base architecture, build "multi-source data analysis, feature extraction, multi-level evidence extraction, active The integrated Chinese and Western medicine big data platform integrates the original evidence processing into a multi-level evidence base, comprehensive analysis of The platform will generate a multi-level evidence base by processing the original evidence, analyze the evaluation indexes of New Coronary Pneumonia, select the features, build a deep neural network model, train and validate the model, and establish a high The model is trained and validated, and a three-level early warning model is established for people at high risk of new coronary pneumonia, those who turn serious, and those with sequelae.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria of mild and moderate types of COVID-19 disease described in the "Diagnostic and Treatment Protocol for Novel Coronavirus Pneumonia (Trial version 9)" [9];
2. Age ≥18 years old and ≤90years old;
3. Not more than 5 days after the occurrence of the first symptom (or confirmed onset);
4. The subject agrees to participate the study and have signed the informed consent form by paper signature, electronic signature of mobile software or voice authorization.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients complicated with severe heart, liver, kidney, blood system and other primary diseases and mental disorders.
3. Patients with disturbance of consciousness, aphasia, dementia and other conditions that prevent them from cooperating with the clinical investigators
4. Patients with incomplete study data.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients
Sampling Method: Non-Probability Sample
Enrollment: 378 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
General Data: | Not more than 5 days after the occurrence of the first symptom (or confirmed onset)
  including age, underlying diseases, body weight, occupation, smoking, alcohol drinking, salt intake and exercise
Environment Indicators: | Not more than 5 days after the occurrence of the first symptom (or confirmed onset)
  air temperature, humidity, and air quality
Auxiliary Examination Indicators: | Not more than 5 days after the occurrence of the first symptom (or confirmed onset)
  blood routine (lymphocyte count, lymphocyte/neutrophil ratio), four coagulation items (PT, APTT, TT, FIB), D-Di, C-reactive protein, erythrocyte sedimentation rate, liver function (ALT, AST, ALP), renal function (BUN, Cr), blood glucose, lung CT
TCM based Evaluation: | Not more than 5 days after the occurrence of the first symptom (or confirmed onset)
  TCM constitution differentiation With reference to the Classification and Determination of Constitutions in TCM issued by the China Association of Traditional Chinese Medicine. There are nine constitution types based on TCM syndrome differentiation

CONTACTS AND LOCATIONS:
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijin, China